CLINICAL TRIAL: NCT02611414
Title: Effectiveness of Transcranial Direct Current Stimulation for the Treatment of Functional Dyspepsia: a Randomized Controlled Trial
Brief Title: Effectiveness of tDCS for the Treatment of Functional Dyspepsia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Ernesto Dornelles (Other)
Responsible Party: Principal Investigator, Carine Leite, Carine Leite, MD, Hospital Ernesto Dornelles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 50793815900005304
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-03

CONDITIONS: Dyspepsia
Keywords: functional dyspepsia; tDCS
MeSH Terms: conditions — Dyspepsia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- anodal tDCS (Experimental): TDCS will be delivered with two saline-soaked sponge electrodes. The main electrode to anodal stimulation will be placed over the motor cortex, M1. The second electrode is neutral and will be placed on the skin overlying the supraorbital region The current will be delivered at the intensity of 2mA for 20 minutes. The procedure will be repeated at five consecutive days.
  Interventions: Device: anodal tDCS
- Sham tDCS (Sham Comparator): Two electrodes are positioned at M1 and supra-orbital área. To deliver sham, the current will be delivered for 30 sec only to elicit tingling skin sensation but no cortical excitability changes. The procedure will be repeated at five consecutive days.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: anodal tDCS — tDCS anodal stimulation over M1 area applied for 20 minutes at five consecutive days.
  Arms: anodal tDCS
Device: Sham tDCS — tDCS sham stimulation over M1 applied for 20 minutes (with current turned off at 30 seconds) at five consecutive days.
  Arms: Sham tDCS

SUMMARY:
Functional dyspepsia is a very common disorder of great challenge to clinical management. A therapeutic targets is up-regulation of visceral pain threshold. The transcranial direct current stimulation (tDCS) is a novel therapy that pursues these properties, besides its safety and easy adherence. There is a great need of new treatments for functional dyspepsia. There is no current study evaluating tDCS for this disease.

DETAILED DESCRIPTION:
Functional dyspepsia is a high prevalent disease with substantial costs to health system. There are many available treatments, but disappointing results are reported in clinical trials.

TDCS is a noninvasive, secure and painless technique of brain stimulation. It is delivered by a battery-operated device that transfers low intensity electrical current to all surface of the brain. Then there is a modulation of cortical excitability and influence on central neurological functions. It has been reported its efficacy for the treatment of many diseases such as depression and chronic pain.

Impairment of central mechanisms of interpretation and threshold of pain are related to functional dyspepsia. Therefore, tDCS may benefit dyspeptic patients.

This study is a double blind randomized controled trial to test tDCS effectiveness on functional dyspepsia. Seventy functional dyspeptic patients will be enrolled, being randomized to either tDCS or sham tDCS.

ELIGIBILITY:
Inclusion Criteria:

* functional dyspeptic patients according to Rome IV criteria
* clinical investigation reporting absence of organic causes of functional dyspepsia

Exclusion Criteria

* history of brain trauma, haemorrhage or ischemia
* implantable devices such as pacemaker
* alcohol or drug abuse
* epilepsy
* severe chronic disease
* non-acceptance to sign up the term of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
PADYQ score | 4 weeks
  Decrease in PADYQ (Porto Alegre Dyspepsia Symptoms Questionnaire) score

SECONDARY OUTCOMES:
HADS score | 4 weeks
  Decrease in HADS score
SF36 score | 4 weeks
  Decrease in SF36 score
Use of drugs for dyspeptic symptoms | 1 and 4 weeks
  Questionnaire about the drugs and number of weekly pills used for symptomatic relief of functional dyspepsia symptoms
Self-reported treatment response | 1 and 4 weeks
  Questionnaire for self-reporting and graduating: worsening/no improvement/improvement after treatment

OTHER OUTCOMES:
Adverse reactions | Daily from day of inclusion until day 5
  A questionnaire to point out if presence of one or more of the 8 previously reported adverse effects of tDCS (such as headache and burning sensation).

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme B Sander, PhD, Principal Investigator — Endoscopy and Gastroenterology Unit Coordinator
Locations (1):
- Hospital Ernesto Dornelles - Endoscopy Unit, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Brunoni AR, Nitsche MA, Bolognini N, Bikson M, Wagner T, Merabet L, Edwards DJ, Valero-Cabre A, Rotenberg A, Pascual-Leone A, Ferrucci R, Priori A, Boggio PS, Fregni F. Clinical research with transcranial direct current stimulation (tDCS): challenges and future directions. Brain Stimul. 2012 Jul;5(3):175-195. doi: 10.1016/j.brs.2011.03.002. Epub 2011 Apr 1. PMID 22037126
- [Background] Ma TT, Yu SY, Li Y, Liang FR, Tian XP, Zheng H, Yan J, Sun GJ, Chang XR, Zhao L, Wu X, Zeng F. Randomised clinical trial: an assessment of acupuncture on specific meridian or specific acupoint vs. sham acupuncture for treating functional dyspepsia. Aliment Pharmacol Ther. 2012 Mar;35(5):552-61. doi: 10.1111/j.1365-2036.2011.04979.x. Epub 2012 Jan 16. PMID 22243034
- [Background] Marlow NM, Bonilha HS, Short EB. Efficacy of transcranial direct current stimulation and repetitive transcranial magnetic stimulation for treating fibromyalgia syndrome: a systematic review. Pain Pract. 2013 Feb;13(2):131-45. doi: 10.1111/j.1533-2500.2012.00562.x. Epub 2012 May 28. PMID 22631436